CLINICAL TRIAL: NCT06034990
Title: ICU Fluid Utilization Survey in Southeast Asia
Acronym: Fluid-SEA
Status: Recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Principal investigator, Chulalongkorn University
Other Study IDs: IRB.457/66
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness
Keywords: Crystalloids; Colloids; Fluid resuscitation; Intensive care unit; Sepsis; Bleeding
MeSH Terms: conditions — Critical Illness; Sepsis; Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survey participants: Participants in this cross-sectional survey will be physicians with specialty in Anesthesiology, Surgery, Critical care medicine, Pulmonology, Nephrology, General Medicine currently working in Surgical or Medical ICU in Southeast Asia in year 2023-2024
  Interventions: Other: 10-min online survey

INTERVENTIONS:
Other: 10-min online survey — This is a cross-sectional study. The data are collected by a 10-min online survey administered to included physicians which will be distributed via online channels such as such as official website or Facebook pages of Society of intensive care or Society of nephrology of corresponding countries.

SUMMARY:
The objective of this study is to examine the use of different types of fluids for resuscitation in different phases of fluid management in 3 types of critically ill patients including (1) not bleeding, not septic but need volume resuscitation (representing normal condition), (2) bleeding but not septic (representing normal vascular integrity but with a loss of intravascular colloids), (3) septic (representing the condition with increase vascular permeability and endothelium damage) in the ICU within Southeast Asia.

The data are collected by a 10-min online survey administered to included physicians which will be distributed via multiple online channels through representatives of each countries.

DETAILED DESCRIPTION:
The objective of this study is to examine the use of different types of fluids for resuscitation in different phases of fluid management in 3 types of critically ill patients including (1) not bleeding, not septic but need volume resuscitation (representing normal condition), (2) bleeding but not septic (representing normal vascular integrity but with a loss of intravascular colloids), (3) septic (representing the condition with increase vascular permeability and endothelium damage) in the ICU within Southeast Asia, and to determine whether co-morbidities with hypoalbuminemia, clinician specialties, hospital practice settings, geographic locations and re-imbursement limitation especially for colloids influence the practice patterns of fluid utilization in different phases in the 3 types of patients. Ultimately, the information provided by this study could also provide basic background information for the design of future clinical trials regarding fluid resuscitation strategies.

The data are collected by a 10-min online survey administered to included physicians which will be distributed via multiple online channels through representatives of each countries.

The survey will start with an inform-consent form prior to starting the survey questions which consist of 13-item questionnaire obtaining information on

1. Demographics data of clinicians taking the survey on primary specialty, region or country of practice and hospital settings.
2. Preferences for volume status indicators.
3. Preferences for fluid resuscitation in 3 types of patients (1. Septic 2. bleeding but not septic 3. not bleeding and not septic) during resuscitation and optimization phase.
4. Preferences for fluid resuscitation in the 3 types of patients with hypoalbuminemia including (1) cirrhosis (2) nephrotic syndrome (3) other significant hypoalbuminemia during resuscitation/optimization phase and stabilization phase
5. The reasons for using colloids for volume expansion
6. The experience of adverse reactions to albumin
7. The awareness and importance of non-oncotic properties of albumin
8. The impact of reimbursement for colloids on resuscitation fluid choice

ELIGIBILITY:
Inclusion Criteria:

1. Specialty must be in Anesthesiology, Surgery, Critical Care Medicine, Pulmonology, Nephrology, Internal Medicine, General Practitioner
2. Practice must be in Southeast Asia hospitals
3. Must work in Surgical ICU, Medical ICU , and/or Mixed ICU

Exclusion Criteria:

1.Physicians who worked in cardiac, neurology or pediatric ICUs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physicians with specialty in Anesthesiology, Surgery, Critical care medicine, Pulmonology, Nephrology, General Medicine currently working in Surgical or Medical ICU in Southeast Asia in year 2023-2024
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Fluid resuscitation practice pattern | 1/9/23-1/9/24
  Preferences for fluid resuscitation in 3 types of patients (1. Septic 2. bleeding but not septic 3. not bleeding and not septic) during resuscitation and optimization phase.

SECONDARY OUTCOMES:
Preferences for volume status indicators. | 1/9/23-1/9/24
  Preferences for volume status indicators and diagnostic tools
Fluid resuscitation practice pattern in hypoalbuminemic state | 1/9/23-1/9/24
  Preferences for fluid resuscitation in the 3 types of patients with hypoalbuminemia including (1) cirrhosis (2) nephrotic syndrome (3) other significant hypoalbuminemia during resuscitation/optimization phase and stabilization phase

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Srisawat, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn university, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller TE, Bunke M, Nisbet P, Brudney CS. Fluid resuscitation practice patterns in intensive care units of the USA: a cross-sectional survey of critical care physicians. Perioper Med (Lond). 2016 Jun 16;5:15. doi: 10.1186/s13741-016-0035-2. eCollection 2016. PMID 27313844